CLINICAL TRIAL: NCT07375355
Title: Explore the Effectiveness and Safety of Scemblix (Asciminib) for Newly Diagnosed CML-CP Patients in China Real World Setting (ASC4CN)
Brief Title: Real-world Study of Scemblix in the Treatment of Chronic Myeloid Leukemia in China
Acronym: ASC4CN
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001J1CN01
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myeloid Leukemia in Chronic Phase
Keywords: CML-CP; Asciminib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study Group: Asciminib treatment

SUMMARY:
This is a multicenter, non-interventional real-world study designed to assess the efficacy and safety of asciminib in patients with newly diagnosed CML.The study uses a prospective data collection design to gather baseline, pre- and post-treatment, and long-term follow-up data, enabling a comprehensive assessment of asciminib's clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all the following criteria:

1. 18 years or older at the time of ICF signing;
2. Newly diagnosed with Ph+ CML-CP within 3 months before enrollment;

   - The diagnosis documentation must include the type and quantitative level of the BCR-ABL1 transcript.
3. Prior treatment with a maximum of 2 weeks of TKIs;
4. Prior treatment with non-TKI regimens, including interferon and hydroxyurea, is allowed;
5. Patients scheduled to initiate treatment with asciminib;

   - Patients beginning asciminib treatment must receive the first dose within 14 days of signing the ICF;
6. Signed ICF.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for inclusion in this study:

1. Previous diagnosis of CML-accelerated phase or blast crisis;
2. Currently participating in an interventional clinical study for CML;
3. Having rare, atypical transcript types that cannot be standardised internationally;
4. Women who are pregnant, lactating or planning to become pregnant during the study;
5. Concurrent other malignancies (refer to the International ICD-11 diagnosis codes, with diagnostic text including carcinoma, malignant neoplasm, etc.);
6. Other conditions that are considered not suitable for the study by the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients newly diagnosed with CML-CP and confirmed with Ph+ CML in medical records
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of MMR | Month 12
  Cumulative rate of major molecular response (MMR) (BCR-ABL1 transcript level ≤ 0.1%) in patients receiving asciminib for 12 months

SECONDARY OUTCOMES:
Cumulative rate of MMR | Month 3, Month 6, Month 9, Month 18 and Month 24
  The cumulative MMR is defined as at least one BCR::ABL1 transcript level ≤ 0.1% during the follow-up period
Cumulative rate of deep molecular response (DMR): MR4 and MR4.5 | Month 3, Month 6, Month 9, Month 12, Month 18, and Month 24
  Cumulative rate of MR4 is defined as at least one BCR::ABL1 transcript level ≤ 0.01% during the follow-up period; Cumulative MR4.5 is defined as at least one BCR::ABL1 transcript level ≤0.0032% during the follow-up period
Cumulative rate of complete cytogenetic response (CCyR) | Month 3, Month 6, and Month 12
  Cumulative CCyR is defined as at least one cytogenetic examination showing 0 Ph+ cells during the follow-up period
Time to first MMR | 24 month follow up period
  Time to first MMR is defined as the time interval from baseline to the first occurrence of BCR::ABL1 transcript level ≤0.1% during the follow-up period
Time to first MR4 and MR4.5 | 24 month follow up period
  Time to first MR4 is defined as the time interval from baseline to the first occurrence of BCR::ABL1 transcript level ≤0.01% during the follow-up period.
  Time to first MR4 is defined as the time interval from baseline to the first occurrence of BCR::ABL1 transcript level ≤0.0032% during the follow-up period
Time to first complete cytogenetic response (CCyR) | 24 month follow up period
  Time to first CCyR is defined as the time interval from baseline to the first occurrence of CCyRduring the follow-up period
Early molecular response (EMR) rate at 3 months | Month 3
  Proportion of patients achieving BCR::ABL1 transcript level ≤10% at M3
Complete hematologic response (CHR) rate | Month 1, Month 2, and Month 3
  the proportion of patients achieving white blood cell count < 10 × 109/L, platelet count < 450 × 109/L, no immature myeloid cells in peripheral blood, peripheral blood basophil percentage < 5%, absence of symptoms/signs of extramedullary involvement, and non-palpable spleen at M1, M2, and M3
Rate of decline in BCR::ABL1 transcript levels | Baseline, Month 1, Month 2, Month 3, Month 6, Month 9 and Month 12
  indirectly calculated from BCR::ABL1 transcript levels at baseline, M1, M2, M3, M6, M9, and M12; determined by BCR::ABL1 halving time
Duration of MMR | 24 month follow up period
  Definition of duration: Duration = sum of "intervals"; Interval calculation method: the first visit at which a response is achieved (and previously unmeasured) within the interval is taken as the starting point, then evaluated sequentially in time order; the calculation stops upon encountering a visit that fails to meet the criterion; The duration is calculated as the time interval between the first and last visit at which the response was achieved; Missing visit data points during this period will be defaulted as achieving the response.
Duration of MR4 and MR4.5 | 24 month follow-up period
Event-Free survival (EFS) rate | Month 12 and Month 24
  Lack of efficacy:
  * Failure to achieve expected molecular response: failure to reach the molecular response milestones recommended by the ELN guidelines at prespecified time points;
  * Loss of molecular response: loss of confirmed MMR following achievement of MMR, or loss of CCyR.
  Disease progression: progression from the chronic phase to the accelerated phase or blast crisis.
  Death: fatal outcome due to any cause during the treatment period. Treatment discontinuation due to adverse events: permanent discontinuation caused by intolerable toxicity, serious adverse events, or other safety-related reasons associated with the study drug.
Progression-free survival (PFS) rate | Month 12 and Month 24
Overall survival (OS) rate | Month 12 and Month 24
Adverse events (AEs) and serious adverse events (SAEs) occurring during asciminib treatment | 24 month follow-up period
Asciminib persistence rates | Month 6, Month 12, and Month 24
Rates of asciminib treatment interruption/dose reduction and discontinuation due to AEs | 24 month follow-up period
Proportion of patients requiring concomitant medications due to AEs | 24 month follow-up period
Change in the simplified CML quality of life questionnaire from baseline | Baseline, Month 12 and Month 24
Compliance following asciminib treatment | 24 month follow-up period
  Medication possession ratio
Concomitant medication use associated with AEs related to asciminib | 24 month follow-up period
Hospitalization rate, outpatient visit rate, emergency department visit rate, and ICU admission rate related to CML treatment | 24 month follow-up period
Gene mutation rate associated with asciminib treatment | 24 month follow-up period
  Gene mutation rate associated with asciminib treatment; types and proportions of positive gene mutations identified via genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No